CLINICAL TRIAL: NCT02663284
Title: Evaluation of Non-invasive Monitor of Physiodoloris Pain in Patients With Complex Regional Pain Syndrome Treated by Nerve Block (Prospective Monocenter Study)
Brief Title: Evaluation of the Physiodoloris Pain Monitor in Patients With Complex Regional Pain Syndrome
Acronym: ANI-ALGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011/67; 2011-A01676-35 (Other: ANSM)
Record Dates: First submitted 2015-09-29; First posted 2016-01-26 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Complex Regional Pain Syndrome
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perineural block (Experimental): Perineural block with Ropivacaine 0.5%
  Interventions: Drug: Ropivacaine 0.5%

INTERVENTIONS:
Drug: Ropivacaine 0.5% — Ropivacaine is used to performed the perineural block

SUMMARY:
A French University team (M. Jeanne, MD, and M. LOGIER, Ph D) have developed a pain assessment tool based on the analysis of the variability heart rate which evaluates the Analgesia Nociception Index (ANI). This index is intended to give a quantification of pain.

The aim of the present study is to assess the validity of the ANI parameter in patients with Complex Regional Pain Syndrome treated with a nerve block (reversible pain).

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from a Complex Regional Pain Syndrome of the upper or lower limb

Exclusion Criteria:

* contra-indication of a nerve block,
* contra-indication of the use of the pain monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of ANI before the peri-neural block | 5 minutes
  ANI is recorded before each nerve block
Evaluation of pain before the peri-neural block | 5 minutes
  Pain score is recorded before each nerve block

SECONDARY OUTCOMES:
Evaluation of ANI after the peri-neural block | 10 minutes
  ANI is recorded after each nerve block
Evaluation of pain after the peri-neural block | 10 minutes
  Pain score is recorded after each nerve block

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, Study Chair — Hopital Foch
Locations (1):
- Clinique des 2 Caps, Coquelles, France